CLINICAL TRIAL: NCT04998214
Title: Hepatic Manifestations and Effect of Long COVID-19 on Patients With Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Huda Mokhtar Salim, clinical professor : Mohammed El _Taher Abdel_Rahman ., Assiut University
Other Study IDs: liver in COVID-19
Record Dates: First submitted 2021-03-19; First posted 2021-08-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Prothrombin Time; International Normalized Ratio

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group non cirrhotic: compare liver function 1m after COVID-19 and that at beginning of infection
  Interventions: Diagnostic Test: liver function , prothrombin time , INR , US .
- cirrhotic patients: compare liver function 1m after COVID-19 and that at beginning of infection
  Interventions: Diagnostic Test: liver function , prothrombin time , INR , US .

INTERVENTIONS:
Diagnostic Test: liver function , prothrombin time , INR , US . — analytic

SUMMARY:
To measure the frequency of persistent liver dysfunction (raised liver enzymes, serum albumin, prothrombin time, etc) in recovered COVID -19 patients.

To compare the hepatic manifestations in post COVID -19 patients with and without liver disease

DETAILED DESCRIPTION:
The digestive tract, particularly the liver, has recently been reported to be affected by SARS-CoV-2. Although abnormal liver enzymes were regularly described as an extra-pulmonary clinical feature, and almost one half of patients experienced grades of hepatic injury. liver damage in patients with SARS infections was primarily manifested in the mild and moderate elevation of alanine and/or aspartate aminotransferases (ALT and AST) with some degree of hypoalbuminemia and hyperbilirubinemia during the early stage of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed by COVID 19 eg : PCR and / or HRCT chest, lab of more than 1 month duration.

Exclusion Criteria:

* Patients less than 18 y.
* Patients with acute COVID 19.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, 1 month post COVID 19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
to evaluate the long term effect of COVID 19 on the liver | 1 month
  to evaluate the changes in liver function (bilirubin ,liver enzymes , albumin , prothrombin time and INR in patients post COVID_19

SECONDARY OUTCOMES:
: Effect of COVID 19 on diseased liver | 1 month
  to evaluate the changes in liver function(bilirubin , liver enzymes , albumin , prothrombin time , INR) in cirrhotic post COVID_19

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Abu Bakr, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Ye ZW, Yuan S, Yuen KS, Fung SY, Chan CP, Jin DY. Zoonotic origins of human coronaviruses. Int J Biol Sci. 2020 Mar 15;16(10):1686-1697. doi: 10.7150/ijbs.45472. eCollection 2020. PMID 32226286
- [Background] Fung SY, Yuen KS, Ye ZW, Chan CP, Jin DY. A tug-of-war between severe acute respiratory syndrome coronavirus 2 and host antiviral defence: lessons from other pathogenic viruses. Emerg Microbes Infect. 2020 Mar 14;9(1):558-570. doi: 10.1080/22221751.2020.1736644. eCollection 2020. PMID 32172672
- [Background] Sultan S, Lim JK, Altayar O, Davitkov P, Feuerstein JD, Siddique SM, Falck-Ytter Y, El-Serag HB; AGA Institute. Electronic address: ewilson@gastro.org. AGA Rapid Recommendations for Gastrointestinal Procedures During the COVID-19 Pandemic. Gastroenterology. 2020 Aug;159(2):739-758.e4. doi: 10.1053/j.gastro.2020.03.072. Epub 2020 Apr 1. No abstract available. PMID 32247018